CLINICAL TRIAL: NCT04515004
Title: Leucoselect Phytosome for Neoadjuvant Treatment of Early Stage Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early termination by sponsor due to substantial delays with subjects recruitment
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONCB-006-19F; I01CX002028 (NIH)
Record Dates: First submitted 2020-08-10; First posted 2020-08-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Early Stage Lung Cancer (I and II)
Keywords: Grape seed procyanidin extract; Early stage lung cancer; Neoadjuvant treatment
MeSH Terms: interventions — leucoselect phytosome

STUDY DESIGN:
Intervention Model Description: This is a phase IIa, single arm study using 2-3 weeks of oral LP treatment for stage I and II lung cancer patients before surgical resection of their tumors
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intervention (Experimental): All qualified participants meeting entry criteria that are enrolled will receive 2-3 weeks of oral LP treatment.
  Interventions: Drug: leucoselect phytosome

INTERVENTIONS:
Drug: leucoselect phytosome — A standardized grape seed procyanidin extract complexed with soy phospholipid.

SUMMARY:
Lung cancer is the leading cause of cancer death in the country, surpassing deaths caused by colorectal, prostate and breast cancers combined. Veterans are at higher risk of lung cancer due to the higher rate of smoking and environmental toxin exposures. The lack of effective therapy for lung cancer provides the impetus to search for alternative, safe, and effective treatment agents to improve treatment strategy against lung cancer, enhance the probability of a cure and reduce recurrence. Based on encouraging preclinical and clinical findings from an early phase I lung cancer prevention study, using a special formulation of a standardized grape seed extract with enhanced absorption called leucoselect phytosome (LP), the purpose of this new CSR&D Merit Review project is to evaluate the potential usefulness of LP for pre-surgical treatment of early stage lung cancer patients in a phase IIa clinical trial. Findings from this study may set the stage for larger, confirmatory trials in the near future.

DETAILED DESCRIPTION:
The investigators will conduct a phase IIa, single arm study using 2-3 weeks of oral LP treatment for 30 early stage I and II lung cancer patients before surgical resection of their tumors.

Screening: Patients who have suspected early stage lung cancer will be recruited from Pulmonary and Thoracic Surgery clinics prior to diagnostic biopsy.

Following informed consent, which includes allowing the investigators to collect and store some of the samples from the clinical diagnostic procedures as pretreatment samples, such as bronchoscopy, needle aspirations, etc., subject will be screened with history and physical examination (H & P), respiratory/general health questionnaires, food frequency self-assessment questionnaires, review of medical records, including radiographic imaging data, pulmonary function test (PFT), 12-lead EKG, clinical labs (complete blood chemistry panel, blood cell counts, PT, PTT). Most of these diagnostic tests will have already been obtained as a part of the clinical work up. However, new blood tests will be obtained if the last results were over 3 months ago). Blood samples and urine samples will be collected for research. Serum cotinine will be obtained to ascertain smoking status. A portion of the biospecimens (blood, urine, diagnostic samples) collected will be kept for future research at the NMVAHCS in an approved repository. A pregnancy test will be done for a woman who is able to have children.

Intervention: (treatment with study medication). If stage I or II lung cancer is diagnosed from standard clinical practice, the qualified subject will be enrolled into the intervention study to receive 2-3 weeks of LP, taken by mouth once a day, until the lung cancer surgery. At the time of surgery, serial clinical samples, including bronchoscopic and various surgically resected tissues, blood and urine will be collected as post-treatment samples. Pre- and post-treatment samples will be compared to assess how well oral LP has been absorbed, and whether or not there are encouraging anti-cancer changes occurring in the cells and molecules in response to the LP treatment. Once enrolled for intervention, all subjects will be monitored with weekly phone follow up, the safety of LP will be monitored weekly using standard reporting tools (including the NCI common terminology criteria for adverse events Version 5.0 and adverse reaction questionnaires), as well as pre-surgery H&P and blood tests.

Follow up: Post-surgery phone follow up will occur at 3-4 weeks, 6 months and annually for up to 4 years.

ELIGIBILITY:
Inclusion Criteria:

A. Initial screening:

* Lesions suspicious for lung cancer
* Competent to provide consent
* CBC within normal limits (WNL)
* liver function test WNL
* Normal Creatinine clearance as measured by the Cockcroft-Gault equation
* ECOG Performance status: 0-1

B. Enrollment for treatment with LP:

* Histologically proven and surgically resectable clinical I and II stage NSCLC

Exclusion Criteria:

* Inability to provide informed consent (e.g. cognitive impairment, severe psychiatric disorders)
* Hypersensitivity to grapes or related products
* Advance respiratory disease (Post resection FEV1 < 0.8 liters, resting hypoxemia, to ensure pts have adequate reserve to undergo diagnostic procedures and surgical resection)
* Unstable angina
* Other concurrent malignancy, excluding non-melanoma type skin cancer
* Have had a solid organ or bone marrow transplant
* Pregnancy
* Breast feeding
* Systemic corticoid steroid therapy of > 10 mg prednisone equivalent daily
* Coagulopathy (PT-INR > 1.2, PTT > 40 seconds) or history of bleeding/clotting problems
* Concurrent use of Grapes or related products
* Unwilling to refrain from drinking more than 1 glass of wine a day
* Pts receiving medications known to be modulators of cytochrome P450 3A4 if alternative medication cannot be provided
* Currently taking other investigational agents
* Pts with concurrent medical conditions that may interfere with completion of tests, therapy, or the follow up schedule

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Delay in the planned surgery of >14 days that is possibly related to study medication (Safety and feasibility). | No greater than 14 days delay in planned surgery.
  Defined as no delay in the planned surgery of >14 days that is possibly related to study medication.

SECONDARY OUTCOMES:
Tumor Ki-67 labeling index (LI), a marker of cell proliferation. | Interim analysis on matched, pre- and post-treatment comparisons will be performed after 10 subjects have completed the treatment portion of the study, anticipated to be in year 2
  Modulations of tumor Ki-67 LI.
Histopathology: pathological response of resected tumor and Lymph nodes. | Interim analysis on matched, pre- and post-treatment comparisons will be performed after 10 subjects have completed the treatment portion of the study, anticipated to be in year 2
  Tumors and lymph nodes with no more than 10% viable tumor cells will be considered to have had a major pathological response.
Tumor activated caspase 3. | Interim analysis on matched, pre- and post-treatment comparisons will be performed after 10 subjects have completed the treatment portion of the study, anticipated to be in year 2
  Modulations of this marker of apoptosis in tumors.

OTHER OUTCOMES:
Tumor COX-2. | Interim analysis on matched, pre- and post-treatment comparisons will be performed after 10 subjects have completed the treatment portion of the study, anticipated to be in year 2
  Modulation of COX-2 expression in Tumor.
15-HETE. | Interim analysis on matched, pre- and post-treatment comparisons will be performed after 10 subjects have completed the treatment portion of the study, anticipated to be in year 2
  Modulations of this marker of inflammation and immunity in biospecimens.
IL-6. | Interim analysis on matched, pre- and post-treatment comparisons will be performed after 10 subjects have completed the treatment portion of the study, anticipated to be in year 2
  Modulations of this marker of inflammation and immunity in biospecimens.
PGE2. | Interim analysis on matched, pre- and post-treatment comparisons will be performed after 10 subjects have completed the treatment portion of the study, anticipated to be in year 2
  Modulations of this marker of inflammation and immunity in biospecimens.
CRP. | Interim analysis on matched, pre- and post-treatment comparisons will be performed after 10 subjects have completed the treatment portion of the study, anticipated to be in year 2
  Modulations of this marker of inflammation and immunity in biospecimens.
MicroRNA (miR)-19a | Interim analysis on matched, pre- and post-treatment comparisons will be performed after 10 subjects have completed the treatment portion of the study, anticipated to be in year 2
  Modulations of this oncogenic miRNA in serum and tumors.
Tumor PTEN. | Interim analysis on matched, pre- and post-treatment comparisons will be performed after 10 subjects have completed the treatment portion of the study, anticipated to be in year 2
  Modulations of this marker of cancerization.
MicroRNA (miR)-19b | Interim analysis on matched, pre- and post-treatment comparisons will be performed after 10 subjects have completed the treatment portion of the study, anticipated to be in year 2
  Modulations of this oncogenic miRNA in serum and tumors.
tumor p-AKT | Interim analysis on matched, pre- and post-treatment comparisons will be performed after 10 subjects have completed the treatment portion of the study, anticipated to be in year 2
  Modulations of this marker of cancerization.
MicroRNA (miR)-106b | Interim analysis on matched, pre- and post-treatment comparisons will be performed after 10 subjects have completed the treatment portion of the study, anticipated to be in year 2
  Modulations of this oncogenic miRNA in serum and tumors.
Stage of lung cancer | Interim analysis on matched, pre- and post-treatment comparisons will be performed after 10 subjects have completed the treatment portion of the study, anticipated to be in year 2
  Change of lung cancer stage based on the American Joint Committee on Cancer (AJCC) TNM staging system.
PGI2. | Interim analysis on matched, pre- and post-treatment comparisons will be performed after 10 subjects have completed the treatment portion of the study, anticipated to be in year 2
  Modulations of this marker of inflammation and immunity in biospecimens.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny T. Mao, MD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/04/NCT04515004/ICF_000.pdf